CLINICAL TRIAL: NCT02317029
Title: A Comparison of Two Biphasic Waveforms and Impact of Oxygen on Myocardial Injury Following Cardioversion
Brief Title: Comparison of Oxygen Interventions and Defibrillator Efficiency
Acronym: CODE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A major adverse event occured (pulsed biphasic waveform arm).
Sponsor: Randers Regional Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 38281
Record Dates: First submitted 2014-03-18; First posted 2014-12-15 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Cardioversion; Cardiac Arrythmias; Myocardial Injury; Defibrillators; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 ("Standard": Oxygen / LIFEPAK 20) (Experimental): 1. Intervention: Cardioversion with a biphasic truncated exponential waveform
  2. Intervention: Hyperoxia during cardioversion
  Interventions: Device: Cardioversion with a biphasic truncated exponential waveform; Procedure: Hyperoxia during cardioversion
- 2 (room air / LIFEPAK 20) (Active Comparator): 1. Intervention: Cardioversion with a biphasic truncated exponential waveform
  2. Intervention: Normoxia during cardioversion
  Interventions: Procedure: Normoxia during cardioversion; Device: Cardioversion with a biphasic truncated exponential waveform
- 3 (Oxygen / Schiller Defigard 5000) (Active Comparator): 1. Intervention: Cardioversion with a pulsed biphasic waveform
  2. Intervention: Hyperoxia during cardioversion
  Interventions: Device: Cardioversion with a pulsed biphasic waveform; Procedure: Hyperoxia during cardioversion
- 4 (Room air / Schiller Defigard 5000) (Active Comparator): 1. Intervention: Cardioversion with a pulsed biphasic waveform
  2. Intervention: Normoxia during cardioversion
  Interventions: Device: Cardioversion with a pulsed biphasic waveform; Procedure: Normoxia during cardioversion

INTERVENTIONS:
Device: Cardioversion with a pulsed biphasic waveform — Cardioversion will be performed by a pulsed biphasic (Multipulse Biowave®) waveform (Schiller Defigard 5000) with an energy setting of 90J, 120J, 150J, 200J. Primary endpoint: The proportion of patients in sinus rhythm four hours post cardioversion.
  Other Names: Schiller Defigard 5000 (SCHILLER AG, Baar, Switzerland)
  Arms: 3 (Oxygen / Schiller Defigard 5000); 4 (Room air / Schiller Defigard 5000)
Procedure: Normoxia during cardioversion — Patients will be treated with room air with a flow of 10-15 L/minute for 3 minutes prior to cardioversion and nasal room air with a flow of 3 L/minute for 30 minutes following cardioversion
  Other Names: room air during cardioversion
  Arms: 2 (room air / LIFEPAK 20); 4 (Room air / Schiller Defigard 5000)
Device: Cardioversion with a biphasic truncated exponential waveform — Cardioversion will be performed by a biphasic truncated exponential waveform (LIFEPAK 20), with a energy setting of 100J, 150J, 200J, 250J. Primary endpoint: The proportion of patients in sinus rhythm four hours post cardioversion.
  Other Names: LIFEPAK 20, Physio Control Inc., Redmond, WA, USA
  Arms: 1 ("Standard": Oxygen / LIFEPAK 20); 2 (room air / LIFEPAK 20)
Procedure: Hyperoxia during cardioversion — Patients will be treated with 100% oxygen with a flow of 10-15 L/minute for 3 minutes prior to cardioversion and nasal 100% oxygen with a flow of 3 L/minute for 30 minutes following cardioversion
  Other Names: 100% oxygen during cardioversion
  Arms: 1 ("Standard": Oxygen / LIFEPAK 20); 3 (Oxygen / Schiller Defigard 5000)

SUMMARY:
Background:

Cardiac arrhythmias can be terminated by electrical current applied by an external defibrillator. This treatment, named cardioversion, has been used for decades in the treatment of atrial fibrillation.

Several kinds of defibrillators exist, though the relative efficacy and safety of these defibrillators is not clear.

During cardioversion, oxygen is being administered, and it has been a long-held belief that oxygen is always beneficial for the patient. This is now being challenged by recent studies suggesting excessive oxygenation to be potentially dangerous for the patients.

Objective:

1. To compare the efficiency and safety of two different defibrillators
2. To investigate the effects of excessive oxygen on injury of the heart following cardioversion.

Experimental design:

Patients will be recruited at the outpatient clinic at the Department of Cardiology, Regional Hospital of Randers, Denmark as a part of the pre-cardioversion check.

Patients will be randomized to cardioversion using one of two defibrillators and randomized to treatment with room air or 100% oxygen.

The cardiac condition will be measured by blood samples before cardioversion, 4 hours after cardioversion and 3 months after cardioversion. Heart rhythm will be measured by ECG before cardioversion, 1 minute-, 30 minutes- and 4 hours after cardioversion.

DETAILED DESCRIPTION:
Background:

Treatment of cardiac arrest includes effective chest compressions, ventilation using high flow oxygen and the delivery of electric shocks (cardioversion). Prompt termination of cardiac arrhythmias and sufficient airway handling including oxygenation are crucial factors for patient outcome. Studies suggest that cardioversion itself may induce myocardial injury; however it is currently unknown whether hyperoxia exacerbate this injury.

Currently, several different biphasic waveforms are in use for cardioversion.The comparative efficacy and safety of these waveforms has not been compared in clinical studies. Commercially available defibrillators use different electrical waveforms that may affect the efficacy of external defibrillation. Although the superiority of biphasic over monophasic waveforms is well established, the relative efficacy and safety of the available biphasic waveforms is not clear.

The long held belief that oxygen (O2) is always beneficial for ill and injured patients is being challenged by recent studies suggesting that excessive oxygenation may result in free-radical mediated tissue damage, resulting in increased morbidity and mortality. Recent guidelines suggest that O2 should be 'titrated' to achieve an appropriate target saturation of 94-98% rather than being administered in an all-or-nothing fashion, particularly in patients with myocardial ischemia or those following resuscitation from cardiac arrest. The Scottish Intercollegiate Guidelines Network (SIGN), British Thoracic Society, National Institute of Health Care Excellence (NICE), European Resuscitation Council and other respected bodies all restrict O2 use to those with hypoxemia, pulmonary oedema or continuing myocardial ischemia, based on expert opinion and pathophysiological reasoning rather than hard evidence.

Studies using patients presenting with shockable life-threatening arrhythmias (e.g. ventricular fibrillation) are difficult to perform for ethical and practical reasons. This study will therefore use patients requiring elective cardioversion for atrial arrhythmias, who are able to give consent and also present a more controlled population. Elective cardioversion is a standard treatment for patients with atrial arrhythmias and is performed as a day case procedure under general anaesthesia.

This study has the following aims:

1. To compare a standard biphasic waveform with a newer pulsed biphasic waveform on which there is little published data
2. To compare the effect of hyperoxia and room air on myocardial injury following cardioversion on which there is no published data.

Methods:

All patients admitted for cardioversion for atrial fibrillation and flutter will be potentially eligible for the study. Patients will be recruited at the Regional Hospital of Randers as a part of the pre-cardioversion check. This is the first contact to patients, and they will receive oral and written information. The oral and written information will be given by a doctor and/or the primary investigator. The information will be given in a quiet setting, and the patients may ask questions about the study. It will be possible for the patient to have a companion present. Informed consent will be obtained from all participants during the pre-cardioversion check or alternatively prior to cardioversion allowing the patient to have a companion present before consent is given. Patients declining to participate in the study will receive treatment according to the standard protocol.

Patients with atrial fibrillation or flutter for ≤48 hours may be cardioverted immediately. Patients with atrial fibrillation or flutter for >48 hours will be required to have a documented weekly international normalized ratio (INR) ≥2.0 (including within 48 hours of cardioversion) or treatment with dabigatranetexilat for three weeks or longer. Alternatively, a transoesophageal echocardiogram documenting absence of intracardiac thrombi is accepted and cardioversion can be performed on treatment with low molecular weight heparin. All patients will be discharged with a recommendation for therapeutic anticoagulation according to current guidelines.

Patient preparation

Patients will be consulted prior to cardioversion; standard blood test will be taken, blood pressure, height and weight will be measured. Information from patient chart (age, gender, morbidity, co-morbidity and medication) will be used to define baseline values. In addition New York Heart Association Functional Classification (NYHA), European Heart Rhythm Association AF-related symptoms (EHRA), American Society of Anaesthesiologists Score (ASA) and Canadian Cardiovascular Society Grading System (CCS) will be recorded during history taking. In addition, information from the patient chart regarding comorbidities, medication etc. will be obtained.

Cardioversion protocol

Blood samples, ECG, blood pressure, oxygen saturation and heart rate will be obtained at baseline and all patients will receive 0.5 mg Rapifen i.v. All patients will be treated with 100 % oxygen or room air, 10-15 L/ minute for 3 minutes before administration of Propofol. All patients will be treated with Propofol 1 mg i.v./kg bodyweight with subsequent 20 mg boluses as needed. Before cardioversion PaO2 will be measured by arterial blood gas (1 mL).

Follow up All patients will be seen at the outpatient clinic after 3 months. Echocardiography will be performed and biomarkers will be measured. Patients will be classified after NYHA, EHRA, ASA and CCS.

Statistics

Regarding waveforms: Assuming the cumulative efficacy, defined as success rate after all delivered shocks, for one of the waveforms is 95%, and for the other waveform ≥80%, a sample size of 75 patients in each group is needed to achieve a power of 80% in rejecting the null hypothesis (that the difference in cumulative efficacy is ≥15%). Continuous variables (number of shocks, delivered energy etc.) are expressed as mean ± SD or median values and compared with Students t-test or equivalent non-parametric test. Categorical variables (e.g. successful cardioversion) are expressed as percentages and compared using the Chi-square or Fisher's exact test (where appropriate). P ≤ 0.05 is considered statistically significant for all comparisons.

Regarding oxygen treatment: It is estimated that 150 patients will be sufficient for the study. After treatment of 60 patients, an interim futility test will be performed. Biomarker data will be analyzed using parametric and non-parametric tests as appropriate. P ≤ 0.05 is considered statistically significant.

Ethics

Approval from The Danish Research Ethics Committee and Danish Data Protection Agency has been obtained. The project will be performed in accordance with the Danish Health Act.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation or -flutter

Exclusion Criteria:

* Patients <18 years of age
* Pregnancy
* Haemodynamically unstable patients
* Other arrhythmias
* Untreated hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Hs-cTnI and Hs-cTnT for room air versus hyperoxia | Change measured from 2 hours before and 4 hours after cardioversion
  High sensitive cardiac Troponin I (Hs-cTnI) and -T (Hs-cTnT) are biomarkers for myocardial injury. Cardiac troponins are measured in plasma as ng/L.
  Change in cardiac troponins (4 hours after cardioversion - pre-cardioversion) will be compared between room air and hyperoxia.
Defibrillator Efficiency: Proportion of patients in sinus rhythm four hours post cardioversion | Heart rhythm measured four hours after cardioversion
  Proportion of patients in sinus rhythm four hours post cardioversion

SECONDARY OUTCOMES:
Cardiac rhythm and change in biomarkers | Biomarkers will be measured within 2 hours before, 4 hours after and 3 months after cardioversion. ECG will be recorded after 1 minute, 30 minutes and four hours after cardioversion.
  Biomarkers will be measured by NT-pro-BNP (ng/L) and Copeptin (pmol/L) at baseline, discharge and at a 3 months follow up visit in the outpatient Clinic. Change in biomarker levels will be compared for patients treated with hyperoxia and room air.
Echocardiography | Performed at baseline, 2-4 hours after and 3 months following cardioversion
  Cardiac function will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Løfgren, MD, PhD, Study Director — Randers Regional Hospital; Kasper G. Lauridsen, MB, Principal Investigator — Randers Regional Hospital; Anders S. Schmidt, MB, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Central Jutland, Denmark

REFERENCES:
- [Derived] Lauridsen KG, Schmidt AS, Adelborg K, Bach L, Hornung N, Jepsen SM, Deakin CD, Rickers H, Lofgren B. Effects of hyperoxia on myocardial injury following cardioversion-A randomized clinical trial. Am Heart J. 2018 Feb;196:97-104. doi: 10.1016/j.ahj.2017.10.006. Epub 2017 Oct 14. PMID 29421020
- [Derived] Schmidt AS, Lauridsen KG, Adelborg K, Torp P, Bach LF, Jepsen SM, Hornung N, Deakin CD, Rickers H, Lofgren B. Cardioversion Efficacy Using Pulsed Biphasic or Biphasic Truncated Exponential Waveforms: A Randomized Clinical Trial. J Am Heart Assoc. 2017 Mar 8;6(3):e004853. doi: 10.1161/JAHA.116.004853. PMID 28275066